CLINICAL TRIAL: NCT04275037
Title: The Hypotensive Effects of Home-Based Isometric Handgrip Training in Older Adults With Pre-Hypertension and Hypertension - The HoldAge Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Institute of Maia (Other)
Collaborators: Aveiro University (Other); Hospital Infante D. Pedro, Centro Hospitalar Do Baixo Vouga (Unknown); Hospital Pedro Hispano, ULS Matosinhos (Unknown); Porto University (Unknown); University of Connecticut (Other); Unidade de Saúde Familiar de Santa Joana (Unknown); Research Center in Sports Sciences, Health Sciences and Human Development (Other); Unidade de Saúde Familiar Serzedelo (Unknown)
Responsible Party: Principal Investigator, Alberto Alves, Assistant Professor, University Institute of Maia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: POCI-01-0145-FEDER-030646
Record Dates: First submitted 2020-02-10; First posted 2020-02-19 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Hypertension; Pre-Hypertension
Keywords: Isometric Handgrip Training; Elderly; Pre-Hypertension; Hypertension
MeSH Terms: conditions — Hypertension; Prehypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Isometric Handgrip Training (Experimental): The 8-week exercise program will include three sessions of isometric handgrip training per week
  Interventions: Other: Isometric Handgrip Training
- Aerobic Exercise Training (Active Comparator): The 8-week exercise program will include three sessions of aerobic exercise per week
  Interventions: Other: Aerobic Exercise Training
- Control Group (No Intervention): The control group will receive usual medical care

INTERVENTIONS:
Other: Isometric Handgrip Training — The 8-week exercise program will include three sessions of isometric handgrip training per week
  Arms: Isometric Handgrip Training
Other: Aerobic Exercise Training — The 8-week exercise program will include three sessions of aerobic exercise per week
  Arms: Aerobic Exercise Training

SUMMARY:
New data suggests that isometric handgrip training (IHT) might become a novel tool in the treatment of hypertension. The main purpose of this research project is to evaluate the effects of home-based IHT on ambulatory blood pressure in older adults with pre-hypertension and hypertension. Eighty-four older adults with pre-hypertension and hypertension will be randomly distributed to one of three groups: home-based IHT, home-based aerobic exercise training (AET), or attention-control group (CON). Each intervention will have a total duration of 8 weeks. At baseline and after completing the intervention, patients will undergo the following evaluations: 24-hour ambulatory blood pressure, cardiorespiratory fitness, endothelial function, damage and repair, arterial stiffness, inflammatory biomarkers, autonomic function, physical activity levels, dietary intake and quality of life. A qualitative analysis will also be applied to enhance the understanding of the efficacy of this intervention from the patient's perspective.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* Secondary Hypertension
* Target Organ Damage
* Coronary Artery Disease
* Heart Failure
* Any Previous Cardiovascular Event
* Peripheral Artery Disease
* Renal Failure
* Chronic Obstructive Pulmonary Disease
* Insulin Dependent Diabetes
* Change of Antihypertensive Medication in the Past 4 Weeks Before Inclusion in the Study
* Smokers
* Those Participating in Regular Physical Activity

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
24h ambulatory blood pressure | Change from baseline to 2 months

SECONDARY OUTCOMES:
Arterial Stiffness | Change from baseline to 2 months
  Assessed by application tonometry using carotid-femoral pulse wave velocity as the gold-standard measure
Endothelial function | Change from baseline to 2 months
  Assessed by brachial artery dilation to endothelial-dependent stimuli using an ultrasound, according to the recommendations
Inflamamtion | Change from baseline to 2 months
  Plasma levels of inflammatory and anti-inflammatory biomarkers including C-reactive protein, Interleukin-10, total nitric oxide and nitrate/nitrite, endothelial Nitric Oxide Synthase
Endothelial cell repair/damage | Change from baseline to 2 months
  Assessed by the circulating number of endothelial progenitor cells and circulating endothelial cells in a peripheral blood by flow cytometry.
Health-related quality of life | Change from baseline to 2 months
  Assessed by the Short-Form 36
Aerobic fitness | Change from baseline to 2 months
  Assessed by Chester Step Test
Weekly physical activity sleep quality | Change from baseline to 2 months
  Measured in seven consecutive days by accelerometry
Intervention quality | two weeks after the intervention
  Assessed by focus group interviews using semi-structured guide with the participants of the experimental groups
Sleep quality | Change from baseline to 2 months
  Measured in seven consecutive days by accelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Alberto J Alves, PhD, Principal Investigator — CIDESD, University Institute of Maia, Maia, Portugal
Locations (10):
- University of Connecticut, Storrs, Connecticut, United States
- Portugal (9):
  - Unidade de Saúde Familiar de Santa Joana, Santa Joana, Aveiro, Aveiro District
  - University Institute of Maia, Maia, Porto District
  - Hypertension Unit, Hospital Pedro Hispano, ULS, Matosinhos, Portugal, Matosinhos Municipality, Porto District
  - Hospital Infante D. Pedro, Centro Hospitalar do Baixo Vouga, Aveiro, Portugal, Aveiro
  - Institute of Biomedicine, Aveiro
  - University of Aveiro, Aveiro
  - Unidade de Saúde Familiar Serzedelo, Guimarães
  - CINTESIS, Faculty of Medicine, Porto, Portugal, Porto
  - Reserach Center in Sports Sciences, Health Sciences and Human Development, Vila Real